CLINICAL TRIAL: NCT05575453
Title: OPTIMA-BP: Empowering PaTients in MAnaging Blood Pressure
Acronym: OPTIMA-BP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INGN21CA393
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
Keywords: Hypertension; Home Blood Pressure Monitoring; Digital health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kvatchii Portal (Active Comparator): The intervention group will be given access to the Kvatchii portal and home blood pressure monitor
  Interventions: Other: Kvatchii Portal
- Usual Care (No Intervention): The control group will not have access to the portal but will be provided with home blood pressure monitor

INTERVENTIONS:
Other: Kvatchii Portal — Online education portal
  Arms: Kvatchii Portal

SUMMARY:
Hypertension is the leading modifiable risk factor for cardiovascular disease and is implicated in half of all strokes and myocardial infarctions. One-third of adults in Scotland have hypertension yet only one-quarter of these have their blood pressure (BP) controlled to target (<140/90 mmHg). Reasons for the low rate of control are varied but include individuals lack of confidence, knowledge and understanding of the condition and treatment strategy, non-adherence to medication and infrequent BP monitoring. These issues have been compounded by the ongoing COVID-19 pandemic which has brought changes in routine BP screening, access to medical care and chronic disease management in primary and secondary care, shielding of the highest risk groups and a change in health and research focus. Shared decision making and issues around health literacy were highlighted by the Scottish Government Cross Party Group on Heart Disease and Stroke: High Blood Pressure Task Force in 2019. Empowering patients to have a better understanding of their condition and becoming actively involved in the monitoring and management of hypertension may lead to improved patient satisfaction, improved BP control and health outcomes and reduction in the use of primary/secondary care hypertension clinics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Current attendance at the GBPC

Exclusion Criteria:

* Inability to give informed consent
* Non-English speakers
* No internet access
* Clinic or ambulatory blood pressure ≥180/120 mmHg
* Arm circumference >42cm
* Inability to perform HBPM
* Inability to use Kvatchii portal
* Pregnancy
* Persistent atrial fibrillation
* Acute cardiovascular event requiring hospitalisation in the previous 3 months
* CKD stage ≥4 or renal dialysis
* Severe or terminal illness limiting study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
HBPM systolic blood pressure (SBP) area under the curve (AUC) | Baseline and 6 months
  HBPM systolic blood pressure (SBP) area under the curve (AUC)

SECONDARY OUTCOMES:
HBPM diastolic blood pressure (DBP) under the curve (AUC) | Baseline and 6 months
  HBPM diastolic blood pressure (DBP) under the curve (AUC)
HBPM systolic blood pressure (SBP) under the curve (AUC) | Baseline and 12 months
  HBPM systolic blood pressure (SBP) under the curve (AUC)
HBPM diastolic blood pressure (DBP) under the curve (AUC) | Baseline and 12 months
  HBPM diastolic blood pressure (DBP) under the curve (AUC)
Change in knowledge of hypertension measured by Blood Pressure Knowledge questionnaire | Baseline, 6 months and 12 months
  True/false questions, 20 items, score 0-20 with higher indicating greater knowledge
Change in health literacy measured by BRIEF: Health literacy Screening Tool | Baseline, 6 months and 12 months
  4 items, score 0-20 with higher score indicating greater health literacy
Change in quality of life measured by EQ-5D-5L questionnaire | Baseline, 6 months and 12 months
  25 items in 5 domains, health state defined by combining one level from each of the 5 domains of the questionnaires. Lower score indicates lower levels of health problems. Visual scale scored out of 100 with higher score indicating better health.
Change in quality of life measured by Patient Health Questionnaire (PHQ-9) questionnaire | Baseline, 6 months and 12 months
  9 items, score 0-27 with higher score indicating greater severity of depression
Change in quality of life measured by the generalised anxiety disorder 7 item scale (GAD-7) | Baseline, 6 months and 12 months
  7 items, score 0-21 with higher score indicating greater anxiety
Change in antihypertensive medicine adherence measured by the Hill-Bone compliance to High Blood Pressure Therapy Scale (HB-HBP) | Baseline, 6 months and 12 months
  14 items, score 0-56 with higher score indicating higher compliance
Change in lifestyle measured by lifestyle questionnaire | Baseline, 6 months and 12 months
  13 items, lower score indicating poorer lifestyle
Antihypertensive medication changes | Baseline, 6 months and 12 months
  Number of antihypertensive medication changes measured by number of medicines altered from last visit
Evaluation of the Kvatchii portal measured by system usability scale (SUS) | over the course of 24 months
  10 items, score 0-100 with higher score indicating better usability

CONTACTS AND LOCATIONS:
Overall Officials: Linsay McCallum, MBChB PhD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Glasgow Clinical Research Facility, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCallum L, Lip S, Rostron M, Hanna R, Bin Pg Md Salimin N, Nichol S, Padmanabhan S. OPTIMA-BP: empOwering PaTients in MAnaging Blood Pressure - protocol for a randomised parallel group study comparing use of Kvatchii web-based patient education portal as an addition to home blood pressure monitoring. Open Heart. 2024 Mar 1;11(1):e002535. doi: 10.1136/openhrt-2023-002535. PMID 38429056